CLINICAL TRIAL: NCT04406454
Title: The Application of Non-invasive and Cellular Level Resolution Fullfield Optical Coherence Tomography: Establishment and Analysis of Subcutaneous Cellular Level Image Database of Anatomical Locations in Healthy Volunteers and Evaluation of Usability
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-01-001A
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Healthy Skin; Nevus
Keywords: Optical Coherence Tomograohy; Healthy volunteer; Non-invasive image system; Cellular level resolution; Full-Field OCT; Nevus
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heathy volunteers: Patients has healthy skin at 5 anatomical locations including face, back, dorsal forearm, volar forearm, calf and at least a nevus without superficial scales and crusting.
  Interventions: Device: ApolloVue® S100 Image System

INTERVENTIONS:
Device: ApolloVue® S100 Image System — The device is an in vivo non-invasive optical coherence tomography and will be used to obtain at least 3 quality OCT images of B-scan (cross-section) and E-scan (en face) with 4 depths for each skin site respectively for each skin site. There is a total of 6 skin sites.

SUMMARY:
ApolloVue® S100 Image System is a medical device class II. The objective of this protocol is to image skin of healthy volunteers and to evaluate the performance of full-field optical coherence tomography (FF-OCT) device - the ApolloVue® S100 Image System in imaging skin microstructures of healthy skin at different anatomical locations and nevi for different skin types and different age and to evaluate usability of the ApolloVue® S100 Image System.

DETAILED DESCRIPTION:
The OCT can provide cellular resolution (~1μm in lateral and axial directions) images. A cellular resolution OCT has the characteristics of non-invasive, non-radioactive, labelfree, real-time and high tissue penetration depth that are highly valuable for clinical use. This technology allows visualization of important structural features such as the epidermis and dermis and the epidermal-dermal junction. OCT has the advantage of generating cross-sectional images, like the orientation of pathology slides.

The ApolloVue® S100 Image System is intended to be used as a non-invasive imaging tool in the evaluation of external human skin tissue microstructure by providing two-dimensional, crosssectional (B-scan) and en face (E-scan) real-time visualization for assessment by physicians to support in forming a clinical judgment. For the ApolloVue® S100 Image System image, both cross-sectional view and en face view can be obtained to assist physicians' diagnosis. With both views, physicians can obtain important spatial information in regards to the skin. Besides, the ApolloVue® S100 Image System is equipped with an image guiding system which provides a high-resolution dermatoscope like image, for the positioning of skin sites for optical biopsies.

In this protocol, it is proposed to study the optical imaging features of healthy human skin and nevi and the evaluation of usability. We propose to recruit 60 subjects for such a trial. Healthy volunteers will be approached and consented to this protocol. The volunteers will be imaged.

ELIGIBILITY:
Inclusion Criteria:

1. All age will be recruited.
2. Both genders will be recruited.
3. All skin types will be recruited. Skin type I-VI (Fitzpatrick scale)

   * Type I always burns, never tans (unexposed skin color: white)
   * Type II usually burns, tans less than average (with difficulty) (unexposed skin color: white)
   * Type III sometimes mild burns, tans about average (unexposed skin color: white)
   * Type IV rarely burns, tans more than average (with easy) (unexposed skin color: white)
   * Type V very rarely burns (unexposed skin color: brown)
   * Type VI never burns (unexposed skin color: black)
4. Has healthy skin at 5 anatomical locations including face, back, dorsal forearm, volar forearm, and calf.
5. Has at least a nevus without superficial scales and crusting
6. Willing to provide informed consent

Exclusion Criteria:

1. Individuals who have a systemic skin disorder.
2. Individuals who have a history of severe skin condition
3. Individuals with surgeries/cosmetic surgeries/micro cosmetic surgery (eg. cosmetic injections and/or laser etc.) on healthy skin at the 5 anatomical locations and nevi (see inclusion criteria 5) in last 12 months and a physician determine the surgery will affect outcome of the OCT images.
4. Not willing to cooperate with methods and related procedures of this trial/study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population from healthy volunteers will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Determine the average scanning success rate of obtaining at least 3 quality OCT images of B-scan and E-scan with 4 depths for each skin site, respectively. | 2 years
  * Scanning efficiency = total number of quality images/total number of images obtained x 100%.
  * Scanning efficiency ≧ 50%
Evaluator identification of each feature will be assessed (number of correctly identified feature/number of total features x 100%). | 2 years
  The purpose of this evaluation is to validate that the ApolloVue® S100 Image System delivers non-invasive skin image features.
  Required features will be analyzed for each group, including age, skin type and anatomical location.
  The features need to meet the following requirement in each 500 x 400 µm2 image for B-scan and in each 500 x 500 μm2 image for E-scan.
  A. Identification of keratinocyte in ≧ 80% of images (B-scan only)
  B. Identification of stratum corneum in ≧ 80% of images
  C. Identification of epidermis in ≧ 80% of images
  D. Identification of dermis in ≧ 80% of images
  E. Identification of EDJ in ≧ 80% of images
  F. Identification of collagen in ≧ 80% of images (B-scan only)
  G. Identification of melanin in ≧ 80% of images
Determine time required to obtain at least 3 quality OCT images of B-scan and E-scan with 4 depths for each skin site, respectively. | 2 years
  Time required < 20 minutes for each body site except for nevus.
  Time required < 40 minutes for a nevus including image guiding.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Dar Lee, M.D., Ph. D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Adabi S, Hosseinzadeh M, Noei S, Conforto S, Daveluy S, Clayton A, Mehregan D, Nasiriavanaki M. Universal in vivo Textural Model for Human Skin based on Optical Coherence Tomograms. Sci Rep. 2017 Dec 20;7(1):17912. doi: 10.1038/s41598-017-17398-8. PMID 29263332